CLINICAL TRIAL: NCT07237165
Title: Evaluation of the Analgesic Effect of Direct Current Stimulation in the Treatment of Pelvic Pain, Comparing Three Groups: Trans-spinal Stimulation, Ganglionic Stimulation, and Placebo. A Randomized Double-blind Study
Acronym: SPINALSTIM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 38RC24.0366
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pelvic Pain
Keywords: Chronic pelvic pain; Non-invasive spinal cord neuromodulation; Trans-spinal direct current stimulation (tsDCS); Trans-spinal stimulation; Dorsal root ganglion stimulation (DRGS)

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trans-spinal stimulation (Active Comparator)
  Interventions: Device: Non-invasive device-based neuromodulation
- Dorsal root ganglion stimulation (Active Comparator)
  Interventions: Device: Non-invasive device-based neuromodulation
- Placebo (non-stimulation (sham) mode) (Placebo Comparator): The device includes a non-stimulation (sham) mode, which can be activated while still placing the electrodes and setting up the device exactly as in the active condition. In this mode, no effective electrical current is delivered, but the procedure appears identical to the real stimulation. This allows the study to maintain double-blind conditions
  Interventions: Device: Non-invasive device-based neuromodulation

INTERVENTIONS:
Device: Non-invasive device-based neuromodulation — Direct current stimulation (tsDCS) protocol consist of one daily session for five consecutive days during the first week, followed by one session per week until week 5, after which the treatment period ends and post-treatment follow-up begins.

SUMMARY:
The purpose of this study is to evaluate the analgesic effectiveness of direct current stimulation (tsDCS) in the treatment of pelvic pain by comparing three groups:

* Trans-spinal tsDCS stimulation,
* Ganglionic tsDCS stimulation,
* Placebo (sham) tsDCS stimulation.

DETAILED DESCRIPTION:
Conduct of study:

Entry into the study: After informed consent, patients will be randomised. The physician responsible for conducting neurostimulation sessions will make the randomization via Redcap. Only this physician will have the knowledge of the group allocated to the patient.

Baseline : Patients, will record on a diary form, a daily Visual Numeric Scale(VNS) of Pain Intensity for 1 week.

Treatment sessions: after the baseline, sessions of neurostimulation will begin for 5 weeks.

After the end of neurostimulation sessions, patients will be followed for 2 weeks.

Throughout their participation in the study, patients will plot on a diary form their daily VNS.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 85 years, suffering from pelvic pain for more than one year (excluding musculoskeletal causes).
* Patient with stable ongoing medication (analgesic or otherwise) for at least one month.
* Patient for whom lack of response to conventional treatments has led the pain specialist or referring physician to consider non-pharmacological therapeutic options.
* Patient reporting a pain intensity score >3 on the Numeric Visual Pain Scale (NVPS) during pre-screening.
* Patient affiliated with the national health insurance system or an equivalent scheme.
* Patient who has provided written informed consent.

Exclusion Criteria:

* History of drug addiction.
* History of psychiatric disorders likely to interfere with the proper conduct of the study.
* Patient with skin lesions in the lumbar region.
* Person unable to understand the study protocol.
* Individuals covered by Articles L1121-5 to L1121-8 of the French Public Health Code, corresponding to all protected persons: pregnant women, women in labor, breastfeeding mothers, individuals deprived of liberty by judicial or administrative decision, or under legal protection.
* Subject currently in the exclusion period of another clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Evolution of Pain | Pain progression will be assessed from week 1 (before treatment) to week 7 (end of treatment)
  Comparison between the 3 groups of the evolution of the weekly value of the Visual Numeric Pain Scale (VNPS): The patient will raise his pain level on a follow-up diary each day. The VNPS average will be calculated for each week. The VNS is a 10-point scale, ranging from 0 (worse) to 10 (better).

SECONDARY OUTCOMES:
Rate of Responding Patients | week 7 compared with baseline
  Patients will be classified as "responders" if they show a reduction in NVPS (Numeric Visual Pain Scale) scores equal to or greater than 30%
Evaluation of the analgesic effect maintenance | Between Week 5 (end of treatment) and Weeks 6 to 7 (post-treatment follow-up).
  Comparison between groups of the daily Numeric Visual Pain Scale (NVPS) values, averaged over 7 days
Assessment of Overall Patient Improvement. | Day 50 from the beginning of tsDCS treatment compared to baseline
  Comparison between the 3 groups of the overall patient improvement using the Clinical Global Impression of Change scale (CGI).The CGI is a 7-point scale, ranging from 1 (better) to 7 (worse).
Quality of Life Improvement. | Day 50 from the beginning of tsDCS stimulation treatment compared to baseline
  Comparison between the 3 groups of the improvement of quality of life using the SF12 (Short Form 12) questionnaire. SF12 includes a mental and social score ranging from 5.89 to 71.97 and a physical score ranging from 9.95 to 70. a high score indicates a better quality of life.
Evolution of Anxiety and Depressive Traits. | Day 50 from the beginning of tsDCS treatment compared to baseline
  Comparison between the 3 groups of the improvement of anxiety and depressive traits using the HADS questionnaire (Hospital Anxiety and Depression Scale).the HADS score varies between 0 and 42. zero corresponding to the best score.
Evolution of Symptomatological Profiles of Neuropathic Pain. | Day 50 from the beginning of tsDCS treatment compared to baseline
  Comparison between the 3 groups of symptomatological profiles of neuropathic pain using NPSI questionnaire (Neuropathic Pain Symptom Inventory).
Sympathetic Autonomic System Injury and Small Fiber Neuropathy. | Day 50 from the beginning of tsDCS treatment compared to baseline.
  Comparison between the 3 groups of sympathetic autonomic system injury and small fiber neuropathy using the Sudoscan® device.
Autonomous System Assessement. | Day 50 from the beginning of tsDCS treatment compared to baseline.
  Comparison between the 3 groups of changes in skin tension and conductance during fMRI examination.
Evolution of the use of analgesic treatments. | From baseline to day 50.
  Comparison between the 3 groups of the evolution of the use of analgesic treatments reported on the diary.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinical Neurophysiology Unit, Henri Mondor University Hospital, Assistance Publique-Hôpitaux de Paris (AP-HP), Créteil, France, Créteil
  - Pain Management Center, Grenoble Alpes University Hospital (CHU Grenoble Alpes), Grenoble

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hodaj H, Payen JF, Lefaucheur JP. A Case of Long-Term Treatment of Chronic Pain Syndrome by Anodal tDCS of the Motor Cortex, Previously Resistant to High-Frequency rTMS and Implanted Spinal Cord Stimulation. Brain Stimul. 2016 Jul-Aug;9(4):618-20. doi: 10.1016/j.brs.2016.02.008. Epub 2016 Mar 22. No abstract available. PMID 27101725
- [Result] Lefaucheur JP, Antal A, Ayache SS, Benninger DH, Brunelin J, Cogiamanian F, Cotelli M, De Ridder D, Ferrucci R, Langguth B, Marangolo P, Mylius V, Nitsche MA, Padberg F, Palm U, Poulet E, Priori A, Rossi S, Schecklmann M, Vanneste S, Ziemann U, Garcia-Larrea L, Paulus W. Evidence-based guidelines on the therapeutic use of transcranial direct current stimulation (tDCS). Clin Neurophysiol. 2017 Jan;128(1):56-92. doi: 10.1016/j.clinph.2016.10.087. Epub 2016 Oct 29. PMID 27866120
- [Result] Hodaj H, Payen JF, Mick G, Vercueil L, Hodaj E, Dumolard A, Noelle B, Delon-Martin C, Lefaucheur JP. Long-term prophylactic efficacy of transcranial direct current stimulation in chronic migraine. A randomised, patient-assessor blinded, sham-controlled trial. Brain Stimul. 2022 Mar-Apr;15(2):441-453. doi: 10.1016/j.brs.2022.02.012. Epub 2022 Feb 25. PMID 35219923
- [Result] Hodaj H, Payen JF, Hodaj E, Dumolard A, Maindet C, Cracowski JL, Delon-Martin C, Lefaucheur JP. Long-term treatment of chronic orofacial, pudendal, and central neuropathic limb pain with repetitive transcranial magnetic stimulation of the motor cortex. Clin Neurophysiol. 2020 Jul;131(7):1423-1432. doi: 10.1016/j.clinph.2020.03.022. Epub 2020 Apr 10. PMID 32387962
- [Result] Hodaj H, Payen JF, Dumolard A, Delon-Martin C, Lefaucheur JP. Treatment of pudendal neuralgia by high-frequency rTMS of the medial wall of motor cortex bilaterally using an angled figure-of-eight coil. Brain Stimul. 2020 Sep-Oct;13(5):1412-1413. doi: 10.1016/j.brs.2020.07.009. Epub 2020 Jul 23. No abstract available. PMID 32712341
- [Result] Hodaj H, Payen JF, Hodaj E, Sorel M, Dumolard A, Vercueil L, Delon-Martin C, Lefaucheur JP. Long-term analgesic effect of trans-spinal direct current stimulation compared to non-invasive motor cortex stimulation in complex regional pain syndrome. Brain Commun. 2023 Jul 1;5(4):fcad191. doi: 10.1093/braincomms/fcad191. eCollection 2023. PMID 37545548
- [Result] Guidetti M, Ferrucci R, Vergari M, Aglieco G, Naci A, Versace S, Pacheco-Barrios K, Giannoni-Luza S, Barbieri S, Priori A, Bocci T. Effects of Transcutaneous Spinal Direct Current Stimulation (tsDCS) in Patients With Chronic Pain: A Clinical and Neurophysiological Study. Front Neurol. 2021 Sep 6;12:695910. doi: 10.3389/fneur.2021.695910. eCollection 2021. PMID 34552550
- [Result] Rahman MA, Tharu NS, Gustin SM, Zheng YP, Alam M. Trans-Spinal Electrical Stimulation Therapy for Functional Rehabilitation after Spinal Cord Injury: Review. J Clin Med. 2022 Mar 11;11(6):1550. doi: 10.3390/jcm11061550. PMID 35329875
- [Result] Fregni F, El-Hagrassy MM, Pacheco-Barrios K, Carvalho S, Leite J, Simis M, Brunelin J, Nakamura-Palacios EM, Marangolo P, Venkatasubramanian G, San-Juan D, Caumo W, Bikson M, Brunoni AR; Neuromodulation Center Working Group. Evidence-Based Guidelines and Secondary Meta-Analysis for the Use of Transcranial Direct Current Stimulation in Neurological and Psychiatric Disorders. Int J Neuropsychopharmacol. 2021 Apr 21;24(4):256-313. doi: 10.1093/ijnp/pyaa051. PMID 32710772
- [Result] Pinto CB, Teixeira Costa B, Duarte D, Fregni F. Transcranial Direct Current Stimulation as a Therapeutic Tool for Chronic Pain. J ECT. 2018 Sep;34(3):e36-e50. doi: 10.1097/YCT.0000000000000518. PMID 29952860
- [Result] Truini A, Vergari M, Biasiotta A, La Cesa S, Gabriele M, Di Stefano G, Cambieri C, Cruccu G, Inghilleri M, Priori A. Transcutaneous spinal direct current stimulation inhibits nociceptive spinal pathway conduction and increases pain tolerance in humans. Eur J Pain. 2011 Nov;15(10):1023-7. doi: 10.1016/j.ejpain.2011.04.009. Epub 2011 May 14. PMID 21576030
- [Result] Cogiamanian F, Vergari M, Pulecchi F, Marceglia S, Priori A. Effect of spinal transcutaneous direct current stimulation on somatosensory evoked potentials in humans. Clin Neurophysiol. 2008 Nov;119(11):2636-40. doi: 10.1016/j.clinph.2008.07.249. Epub 2008 Sep 10. PMID 18786856
- [Result] Priori A, Ciocca M, Parazzini M, Vergari M, Ferrucci R. Transcranial cerebellar direct current stimulation and transcutaneous spinal cord direct current stimulation as innovative tools for neuroscientists. J Physiol. 2014 Aug 15;592(16):3345-69. doi: 10.1113/jphysiol.2013.270280. Epub 2014 Jun 6. PMID 24907311
- [Result] Cogiamanian F, Ardolino G, Vergari M, Ferrucci R, Ciocca M, Scelzo E, Barbieri S, Priori A. Transcutaneous spinal direct current stimulation. Front Psychiatry. 2012 Jul 4;3:63. doi: 10.3389/fpsyt.2012.00063. eCollection 2012. PMID 22783208
- [Result] Nitsche MA, Paulus W. Sustained excitability elevations induced by transcranial DC motor cortex stimulation in humans. Neurology. 2001 Nov 27;57(10):1899-901. doi: 10.1212/wnl.57.10.1899. PMID 11723286
- [Result] Nitsche MA, Liebetanz D, Lang N, Antal A, Tergau F, Paulus W. Safety criteria for transcranial direct current stimulation (tDCS) in humans. Clin Neurophysiol. 2003 Nov;114(11):2220-2; author reply 2222-3. doi: 10.1016/s1388-2457(03)00235-9. No abstract available. PMID 14580622
- [Result] Medeiros LF, de Souza IC, Vidor LP, de Souza A, Deitos A, Volz MS, Fregni F, Caumo W, Torres IL. Neurobiological effects of transcranial direct current stimulation: a review. Front Psychiatry. 2012 Dec 28;3:110. doi: 10.3389/fpsyt.2012.00110. eCollection 2012. PMID 23293607
- [Result] Margueritte F. Algies pelviennes chroniques : prévalence et caractéristiques associées dans la cohorte Constances. Revue d'Epidémiologie et de Santé Publique 2016, Doi : 10.1016/j.respe.2016.01.094
- [Result] Rahman A, Reato D, Arlotti M, Gasca F, Datta A, Parra LC, Bikson M. Cellular effects of acute direct current stimulation: somatic and synaptic terminal effects. J Physiol. 2013 May 15;591(10):2563-78. doi: 10.1113/jphysiol.2012.247171. Epub 2013 Mar 11. PMID 23478132